CLINICAL TRIAL: NCT06183697
Title: Clinical Study for Multi-omics Database Construction of a Cohort of Healthy Korean Volunteers for Integrative Microbiome Analysis
Brief Title: Multi-omics Database Construction of Healthy Korean Volunteers
Status: Recruiting | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, BoHyung Kim, Professor, Kyunghee University Medical Center
Other Study IDs: MB-HV-01
Record Dates: First submitted 2023-11-23; First posted 2023-12-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this prospective, observational study is to collect health-related data including microbiome, blood samples, and dietary habits from the oral and gastrointestinal tracts in healthy subjects. In addition, the study aims to perform microbiome and multi-omics analysis on the collected samples and build an integrated database of the data.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 13 years old and no older than 85 years old at the time of giving their informed consent.
* Subjects who have received a comprehensive explanation of this study, fully understand it, and have voluntarily agreed to participate, providing signed and dated informed consent.
* Subjects considered eligible for participation in the study by the researcher, based on screening procedures including physical examination, clinical laboratory tests, and questionnaires.

Exclusion Criteria:

* Subjects with a Body Mass Index (BMI) below 17.0 or above 30.0.
* Vital signs at rest showing a systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg, along with symptoms related to high blood pressure such as headaches.
* History of using specified drugs within a predetermined period before microbiome collection, as detailed in the Appendix.
* Receipt of any vaccination within the last 4 weeks prior to microbiome collection.
* Use of topical antibiotics or steroids on the face, scalp, neck, arms, forearms, or hands within 24 hours before microbiome collection.
* Application of vaginal or vulvar medications, including antifungals, within 24 hours of microbiome collection.
* Presence of an acute disease at the time of enrollment. Acute disease is defined as the presence of a moderate or severe illness with or without fever. Sampling can be deferred until the subject recovers.
* History of chronic, clinically significant disorders affecting the hepatic, digestive, circulatory, renal, neurological, respiratory, endocrine, immune, or hematological systems, as well as malignant tumors, psychiatric conditions, or substance abuse.
* Substantial dietary alterations for rapid weight gain or loss within 4 weeks of the microbiome collection.
* Positive serological tests (HBs antigen, HCV antibody, and HIV antibody tests) or results above the reference range.
* History of gastrointestinal surgery, excluding simple procedures like appendectomy, cholecystectomy, or hernia repair.
* Presence of gastrointestinal conditions that may influence microbiome analysis and are not under medical control, including Inflammatory Bowel Disease (IBD) including Crohn's disease and ulcerative colitis, Irritable Bowel Syndrome (IBS) requiring medication, ulcers, acute or chronic pancreatitis, and chronic constipation requiring medication.
* Diagnosis of ankylosing spondylitis.
* Requirement for the regular use of incontinence diapers.
* Positive pregnancy test, or being pregnant or lactating.
* Any medical condition suspected at the time of microbiome collection that may affect the integrity of the sample.

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Relative abundance of microbome | 5 years
  Analysis of the microbial community composition will be performed using 16s rRNA gene amplicon sequencing. The relative abundance of microbial species at the genus or family level will be assessed.
Alpha diversity of microbiome (Shannon diversity index) | 5 years
  Alpha diversity will be measured using Shannon diversity index to combine ASV richness and abundance into a single evenness value
Alpha diversity of microbiome (Fisher's index) | 5 years
  Alpha diversity will be measured using Fisher's index, which calculates the relationship between abundance and number
Alpha diversity of microbiome (Faith's phylogenetic diversity whole tree) | 5 years
  Alpha diversity will be measured using Faith's phylogenetic diversity whole tree, representing the sum of all branch lengths as a measure of phylogeny and diversity.

SECONDARY OUTCOMES:
Gene count (transcriptomics) | 5 years
  Analysis of bacterial mRNA profiles will be performed through read mapping using NCBI RefSeq database, quantification of gene and transcript & bacterial taxonomic profiling using HUMAnN and MetaPhlAn pipeline, transcript quantification and identification of differentially expressed gene using SALMON and human reference genome fastq file.
Metabolite peak area (metabolomics) | 5 years
  Analysis of metabolites will be performed by matching metabolite ID achieved from LC/MS with Human Metabolome Database (HMDB) for metabolite identification. Analysis on the difference of metabolite between groups will be performed by PCA or PLS-DA using MZmine3, OpenChrome or Metaboanalyst v5.0.
Relative abundance (virome) | 5 years
  Analysis of total virus profiles will be performed by comparing viral protein sequence with NCBI refseq viral database and taxonomy annotation.
Number of differentially abundant bacterial strains isolated (culturomics) | 5 years
  Bacterial strains that exhibit differential abundance between healthy individuals and patients will be inoculated, isolated, and identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HS, Kim BH, Nam B, Oh SJ, Park SK, Lee SW, Lee JY, Jo S, Lee YA, Lee JY, Park DI, Kim TH, Lee CK. Oral-gut microbiome axis in a Korean cohort with inflammatory bowel disease and ankylosing spondylitis (INTEGRATE): a prospective and observational study protocol. BMJ Open. 2025 Aug 10;15(8):e092075. doi: 10.1136/bmjopen-2024-092075. PMID 40784769